CLINICAL TRIAL: NCT05909176
Title: Start the Conversation: Evaluating Implementation of a Multi-level PrEP Initiative for Black Cisgender Women in New Orleans, Louisiana
Brief Title: Start the Conversation: Evaluating Implementation of a Multi-level PrEP Initiative for Black Cisgender Women in Nola
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO00113159; R34MH129211 (NIH)
Record Dates: First submitted 2023-05-23; First posted 2023-06-18 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2024-12

CONDITIONS: Preexposure Prophylaxis; HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Start the Conversation Package (Experimental): The pre-intervention phase will last for 4 months (months 1-4). The only study activity during the pre-intervention phase is the collection of routine PrEP uptake data to establish a baseline for PrEP prescribing at the GYN residency clinics and local PrEP clinics. The implementation of the combined-care model at the LSU GYN residency clinic at UMCNO for 10 months (months 5-14). Then we will add implementation of the social media campaign in the NOLA area for 4 months (months 5-18); implementation of the combined-care model at LSU GYN residency clinic at UMCNO will continue. The layered approach allows for an opportunity to assess the effect of the combined-care model, and subsequently, to what extent the social media campaign additionally engages Black women and builds demand for PrEP.
  Interventions: Behavioral: GYN Residency Training; Behavioral: Social Media Campaign

INTERVENTIONS:
Behavioral: GYN Residency Training — The combined care model will be implemented and during months 5-14.
Behavioral: Social Media Campaign — The social media campaign will be implemented along with the combined care model in months 15-18.

SUMMARY:
The study objectives are to:

* Evaluate implementation outcomes from piloting the Start the Conversation Initiative
* Assess initial indicators of clinical effectiveness among patients engaged in the Start the Conversation Initiative

These outcomes will be assessed qualitatively through in-depth interviews (IDIs), debriefing sessions with GYN residents and leadership, medical chart reviews and/or de-identified Epic queries, training records, discussions with the Black Women and PrEP (BWAP) Task Force, and social media metrics.

ELIGIBILITY:
Inclusion Criteria:

* LSU GYN residents
* Black cisgender women eligible for PrEP per CDC guidelines

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Total number of women overall and number of Black cisgender women with whom GYN residents start the conversation about PrEP. | Up to 12 months
Total number of women overall and number of Black cisgender women initiating PrEP at the LSU GYN clinic during the pre-implementation period compared to during the two implementation period phases. | Up to 12 months
Comparison of the difference in patient numbers at the LSU GYN clinic during pre-implementation and the two implementation period phases with the difference in patient numbers during the same time frame at the Tulane GYN clinic. | Up to 12 months
Number of patients seen at LSU GYN clinic & UMC PrEP clinic combined compared to the number of patients seen at Tulane GYN & PrEP clinics combined | Up to 12 months

SECONDARY OUTCOMES:
Proportion of PrEP-eligible women overall and Black cisgender women initiating PrEP at the LSU GYN clinic across the two implementation time periods: care model plus social media campaign. | Up to 12 months
Proportion of women choosing follow-up care at the LSU GYN resident clinic versus transition to a local PrEP provider. | Up to 12 months
Proportion of women initiating PrEP at the LSU resident GYN clinic who complete their first follow-up PrEP care visit (can only assess at the LSU GYN resident clinic or UMC PrEP clinic). | Up to 12 months
Number of contacts with the LDH navigator | Up to 12 months
Number of appointments made through the LDH navigator | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Amy Corneli, MPH, PhD, Principal Investigator — Duke University; Meredith Clement, MD, Principal Investigator — Louisiana State University Health Sciences Center
Locations (1):
- Louisiana State University Health Sciences Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing during study implementation: Implementation outcomes will be fed back in real-time to the gynecology residents and the Training Director to inform the residents of implementation fidelity and gain feedback into strategy adaptation. Data sharing will thus be part of the quality improvement process for providers.
  Data sharing after study implementation: Within two months of publication of any manuscript presenting major study findings, study investigators will make the study data available upon request. For the qualitative data, given its descriptive nature, sharing individual transcripts could potentially identify a participant. We will therefore provide de-identified, aggregated data summaries. De-identified implementation outcome data will be made available upon request following publication; we will ensure that data cannot be used to determine resident provider identities or patients.
  Our research will not produce patentable products or involve model organisms.

DOCUMENTS (1):
  • Study Protocol (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT05909176/Prot_000.pdf